CLINICAL TRIAL: NCT03900819
Title: Evaluation of Manual Dexterity in a Monocentric Cohort of Peritoneal Dialysis Patients
Brief Title: Evaluation of Dexterity in Prevalent Peritoneal Dialysis Patients
Acronym: DEXTER
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A01523-52
Record Dates: First submitted 2018-09-20; First posted 2019-04-03 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Peritoneal Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dexterity measurement — 4 non-invasive tests will be performed

SUMMARY:
The objective of the study is to measure the manual dexterity of patients treated by peritoneal dialysis - transversal study

DETAILED DESCRIPTION:
All peritoneal dialysis patients from Peritoneal Dialysis unit will, after information and consent, have to realise four tests, one time each, to quantify their manual dexterity. The tests are already used to measure dexterity: Purdue Pegboard, Jebsen test, JAMAR, Pinch test. These tests will be performed during an in-hospital visit.

ELIGIBILITY:
Inclusion Criteria:

* patients treated by peritoneal dialysis in Caen University Hospital

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All prevalent PD patients from our center will be included
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
success of dexterity measurement in peritoneal dialysis patients evaluated by the Purdue Pegboard | baseline
  number of completed tests (Purdue Pegboard - number inserted in 30 second)
success of dexterity measurement in peritoneal dialysis patients evaluated by the Jebsen test | baseline
  number of completed tests (Jebsen test - time in second)
success of dexterity measurement in peritoneal dialysis patients evaluated by the JAMAR | baseline
  number of completed tests (JAMAR - in kilogramms)
success of dexterity measurement in peritoneal dialysis patients evaluated by the Pinch test | baseline
  number of completed tests (Pinch testin - kilogramms)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided